CLINICAL TRIAL: NCT00664599
Title: Effect of Rituximab in the Treatment of Resistant Ocular Inflammatory Lesions of Behcet's Disease (Pilot Study)
Brief Title: Rituximab for the Treatment of Severe Ocular Manifestations of Behcet's Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Tehran University of Medical Sciences (Other)
Collaborators: Hoffmann-La Roche (Industry)
Responsible Party: Fereydoun Davatchi, Head Rheumatology Research Center, Rheumatology Research Center, Tehran University for Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 132/12487
Record Dates: First submitted 2008-04-20; First posted 2008-04-23 (Estimated); Last update posted 2008-04-30 (Estimated); Status verified 2008-04

CONDITIONS: Behcet's Syndrome
Keywords: Ocular lesions, Visual Acuity, Retinal Vasculitis
MeSH Terms: conditions — Behcet Syndrome; Retinal Vasculitis | interventions — Rituximab; Cyclophosphamide

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Rituximab
  Interventions: Drug: Rituximab
- 2 (Active Comparator): Cytotoxics combination
  Interventions: Drug: Cytotoxic Combination

INTERVENTIONS:
Drug: Rituximab — Infusion of Rituximab, 1500 mg, two times with 15 days interval. Patients receive also Methotrexate (15 mg weekly) and Prednisolone (0.5 mg/daily).
  Other Names: Mabthera; Rituxan
  Arms: 1
Drug: Cytotoxic Combination — Pulse cyclophosphamide 1000 mg in perfusion, once monthly monthly. Azathioprine 3 mg/kg/body weight daily + prednisolone 0.5 mg/kg/daily.
  Other Names: Cytoxan
  Arms: 2

SUMMARY:
The purpose of this study is to find if Rituximab can improve severe ocular lesions of Behcet's Disease.

DETAILED DESCRIPTION:
To test in a single blind randomized control study the efficacy of Rituximab versus combination of pulse cyclophosphamide and azathioprine. Both group receiving 0.5 mg/kg/daily prednisolone.

ELIGIBILITY:
Inclusion Criteria:

* Behcet's Disease fulfilling the new International Criteria for Behcet's Disease
* Having active ocular lesions (posterior and/or retinal vasculitis)
* Resistant to cytotoxic drugs + prednisolone 0.5 mg/kg

Exclusion Criteria:

* Visual acuity less than 1/10 on Snellen chart
* Antecedent of allergic reaction to any component of the therapeutic regimen

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2006-04; Primary Completion 2008-01 (Actual); Study Completion 2008-01 (Actual)

PRIMARY OUTCOMES:
Visual acuity | 6 months

SECONDARY OUTCOMES:
Inflammatory index for posterior uveitis | 6 months
Inflammatory index for retinal vasculitis, especially for edema | 6 months
Total Adjusted Disease Activity Index (TADAI) | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Fereydoun Davatchi, MD, Study Chair — Rheumatology Research Center, Tehran University for Medical Sciences; Hormoz Shams, MD, Principal Investigator — Rheumatology Research Center, Tehran University for Medical Sciences; Mozhgan Rezaipoor, MD, Principal Investigator — Rheumatology Research Center, Tehran University for Medical Sciences; Farhad Shahram, MD, Principal Investigator — Rheumatology Research Center, Tehran University for Medical Sciences; Cheyda Chams-Davatchi, MD, Principal Investigator — Rheumatology Research Center, Tehran University for Medical Sciences; Bahar Sadeghi, MD, Principal Investigator — Rheumatology Research Center, Tehran University for Medical Sciences
Locations (1):
- Rheumatology Research Center, Shariati Hospital, Tehran, Tehran Province, Iran